CLINICAL TRIAL: NCT04741477
Title: The Pharmacokinetics and Pharmacodynamics of Hemp-based Topical Cannabinoid Products
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00277556; 1-340-0216610-65527L (Other Grant/Funding Number: Substance Abuse And Mental Health Administration)
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Cannabis; Drug Effect
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: A total of 5 topical cannabinoid products will be examined in this study. The study will be conducted in 5 discrete stages, one for each product. In each stage, participants (N=20), will be randomized to 1 of 2 double-blind drug conditions that entail the use of: 1) a topical product that contains CBD and a low amount of THC (N=15), or 2) a placebo topical product that does not contain cannabinoids (N=5), but which contains similar non-cannabinoid ingredients to the active product.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topical CBD Product with low level of THC (Experimental): Participants will topically apply a high CBD-product that also contains low levels of THC.
  Interventions: Drug: CBD; Drug: THC
- Placebo topical product (Placebo Comparator): Participants will topically apply a placebo product that does not contain cannabinoids.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBD — CBD will be topically applied
  Arms: Topical CBD Product with low level of THC
Drug: THC — THC will be topically applied
  Arms: Topical CBD Product with low level of THC
Drug: Placebo — a placebo product (without cannabinoids) will be topically applied
  Arms: Placebo topical product

SUMMARY:
This study will evaluate the pharmacokinetic and pharmacodynamic effects of hemp-based Cannabidiol (CBD) topical products (e.g., lotions, creams, patches) that contain low levels of delta-9-tetrahydrocannabinol (THC).

DETAILED DESCRIPTION:
A total of 5 topical cannabinoid products will be examined in this study. The study will be conducted in 5 discrete stages, one for each product. In each stage, participants (N=20), will be randomized to 1 of 2 double-blind drug conditions that entail the use of: 1) a topical product that contains CBD and a low amount of THC (N=15), or 2) a placebo topical product that does not contain cannabinoids (N=5), but which contains similar non-cannabinoid ingredients to the active product. Thus, overall 100 participants will complete the study (75 active, 25 placebo).

Participants in each stage will complete a three-phase outpatient protocol that will last a total of 17 days. Phase 1 (Day 1) will be an acute laboratory dosing session (approximately 7 hours in duration). Phase 2 (Days 2-10) will be an outpatient dosing period, during which participants will continue to use participants' assigned product twice daily (morning and evening) in participants' own environment. During Phase 2, participants will visit the laboratory for brief study sessions on Days 2, 3, 7, and 10. Phase 3, will consist of a final follow-up visit on Day 17, after a 1-week drug washout. Pharmacokinetic and pharmacodynamic assessments (subjective and cognitive effects) will be assessed during each phase.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Be between the ages of 18 and 55
3. Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
4. Test negative for recent cannabis use in urine at the screening visit and again upon admission for each experimental session
5. Test negative for other drugs of abuse, including alcohol, at the screening visit and upon arrival for each experimental session
6. Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at each study visit.
7. Have a body mass index (BMI) in the range of 19 to 36 kg/m^2
8. Have head hair that is at least 4 cm (approximately one and a half inches) in length on the back of the head.
9. Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
10. Report prior experience using cannabis or CBD products.
11. Have not donated blood in the prior 30 days.
12. Have a smart phone, tablet, computer, etc. capable of recording videos and operating Redcap.

Exclusion Criteria:

1. Non-medical use of psychoactive drugs other than, nicotine, alcohol, or caffeine in the month prior to the screening visit.
2. History of or current evidence of significant medical or psychiatric illness judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
3. Use of an over-the-counter (OTC), systemic or topical drug(s), herbal supplement(s), vitamin(s), or prescription medications (with the exception of birth control prescriptions) within 14 days of study entry; which, in the opinion of the investigator or sponsor, will interfere with the study results or the safety of the subject.
4. Use of hemp seeds or hemp oil in any form in the past 3 months.
5. Use of dronabinol (Marinol) within the past 6 months.
6. History of xerostomia (dry mouth), or the presence of mucositis, gum infection or bleeding, or other significant oral cavity disease or disorder that in the investigator's opinion may affect the collection of oral fluid samples.
7. History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
8. Known allergy to any ingredients in the active or placebo topical products.
9. Enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing.
10. Epilepsy or a history of seizures.
11. Individuals with anemia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Change in Urine cannabinoids | Days 1, 2, 3, 7, 10, and 17
  Concentration of cannabinoids will be measured in urine (unit of measurement: nanograms/mL)
Change in Blood cannabinoids | Days 1, 2, 3, 7, 10, and 17
  Concentration of cannabinoids will be measured in blood (unit of measurement: nanograms/mL)

SECONDARY OUTCOMES:
Change in Oral fluid cannabinoids | Days 1, 2, 3, 7, 10, and 17
  Concentration of cannabinoids will be measured in oral fluid (unit of measurement: nanograms/mL)
Change in Hair cannabinoids | Days 1 and 17
  Concentration of cannabinoids will be measured in hair (unit of measurement: nanograms/mL)
Change in Subjective drug effects as assessed by the Drug Effect Questionnaire | Days 1, 2, 3, 7, 10, and 17
  Subjective drug effect ratings (0-100) will be collected with the Drug Effect Questionnaire, with 0 being no effect and 100 being maximum effect.
Change in Cognitive performance as assessed by the Divided Attention Task | Days 1, 2, 3, 7, 10, and 17
  Cognitive performance will be evaluated with the Divided Attention Task. Will be measured as the mean distance (in computer pixels) of the mouse cursor from the central stimulus.
Change in Working memory performance as assessed by the Paced Serial Addition Task | Days 1, 2, 3, 7, 10, and 17
  Working memory performance will be evaluated with the Paced Serial Addition Task (scores can range from 0-90) with 90 indicating perfect performance.
Change in Psychomotor performance as assessed by the Digit Symbol Substitution Task | Days 1, 2, 3, 7, 10, and 17
  Psychomotor performance will be evaluated with the Digit Symbol Substitution Task. Will be measured as the number of correct trials within 90 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Tory Spindle, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No